CLINICAL TRIAL: NCT06553352
Title: An Open, Single-Arm Clinical Study of Zanubrutinib in Combination With Obinutuzumab (ZO) for Newly Diagnosed Follicular Lymphoma (FL)
Brief Title: Zanubrutinib in Combination With Obinutuzumab (ZO) for Newly Diagnosed Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: Shanxi Provincial Cancer Hospital (Unknown); The First Hospital of Jilin University (Other); Fujian Cancer Hospital (Other Government); Jiangxi Provincial Cancer Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Sun Yat-sen University (Other); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-10
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Follicular Lymphoma; Newly Diagnosed
MeSH Terms: conditions — Lymphoma, Follicular | interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Z) combined with Obinutuzumab (O) (Experimental): Zanubrutinib (Z) 160mg bid oral d1-21 Obinutuzumab (O) C1 1000mg d1,8,15 C2-C6 d1 IV, then every 8 weeks until full 20 infusions (1 years maintenance)
  Interventions: Drug: Zanubrutinib combined with Obinutuzumab

INTERVENTIONS:
Drug: Zanubrutinib combined with Obinutuzumab — Zanubrutinib combined with Obinutuzumab (ZO), a specific dose on specific days.
  Other Names: Zanubrutinib combined with Obinutuzumab (ZO)

SUMMARY:
To evaluate the efficacy and side effects of Zanubrutinib combined with Obinutuzumab (ZO) in the treatment of newly diagnosed follicular lymphoma.

DETAILED DESCRIPTION:
Zanubrutinib (Z) 160mg bid oral d1-21 Obinutuzumab (O) C1 1000mg d1,8,15 C2-C6 d1 IV, then every 8 weeks until full 20 infusions (1 year maintenance)

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old and gender-neutral;
2. Follicular lymphoma definitively diagnosed according to the REAL/WHO classification, stage II-IV requiring treatment according to the GELF code;
3. ECOG score 0-2;
4. Lymphoma efficacy evaluation criteria using Lugano 2014 Lymphoma must have at least one measurable or evaluable lesion: signed informed consent, subjects recruited based on inclusion and exclusion criteria, etc History taking and pre-treatment baseline examination and registration on case report form (CRF) ZO regimen of chemotherapy for 6 cycles, followed by zebrutinib monotherapy orally for 6 months, with observation of toxicities Follow-up assessment (including) Follow-up evaluation (including safety) <Blood, biochemistry, B2-MG, neck, chest and abdomen CT plain + enhanced, questionnaire> Follow-up evaluation (including safety) <Blood, biochemistry, B2-MG, neck, chest and abdomen CT plain + enhanced, questionnaire, once every three months> 1. Zerbutinib maintenance treatment for 12 months for PR and above 2. Second-line treatment for the rest of the patients (recommended by NCCN guidelines) NCCN guideline recommendation) Assessment of efficacy i.e. PET/CT with evaluable lesions; CT or MR evaluation of intranodal lesions with a long diameter >1.5cm, short diameter >1.0cm or extranodal lesions with a long diameter >1.0cm;
5. HBV-positive serology (concealed carriers: anti-HBeAg +, HbsAg-, anti-HBsAg +/-) Enrollment only if HBV-DNA test is negative;
6. Normal major organ function: liver function serum bilirubin ≤ 2.0 × ULN , serum ALT and AST ≤ 2.5 × ULN, renal function: serum Cr ≤ 2.0 × ULN; (unless due to lymphoma);
7. Informed consent (patients must sign an informed consent form for all studies).

Exclusion Criteria:

1. Medically significant CNS lymphoma or molluscum contagiosum or large cell transformation;
2. HIV-positive patients and or HCV active infection (documented by HCV-RNA positive test);
3. Patients should not have active or uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia Patients should not have transfusion-dependent thrombocytopenia or bleeding disorders Patients should not have autoimmune disorders associated with the study drug;
4. Known bleeding disorders (e.g., vascular hemophilia or hemophilia) in combination with warfarin or other vitamin K antagonists require treatment with a potent cytochrome P450 (CYP) 3A inhibitor;
5. Patients with acute coronary syndrome within 6 months prior to study entry must not have had a stroke or intracranial hemorrhage within the past 6 months Prior Surgery: no major surgery within 28 days prior to enrollment or minor surgery within 7 days prior to enrollment; examples of minor surgery include dental procedures, venous access device insertion, skin biopsies, or joint aspirations; procedures may be major or minor at the discretion of the treating physician;
6. Severe COPD with combined hypoxemia;
7. Active bacterial, fungal, and, or viral infections not controlled by systemic therapy;
8. In addition to cured basal cell carcinoma of the skin or cervical cancer in situ or early prostate cancer that does not require systemic therapy, or early breast cancer that requires surgery alone. Other malignant tumors within the last 2 years or concurrently;
9. Pregnancy and Lactation: Female patients must have a negative serum pregnancy test within 72 hours prior to initiation of regimen therapy and use effective contraception during regimen therapy and for at least 12 weeks after completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
CR | up to 1 year
  Complete remission rate

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- Bing Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided